CLINICAL TRIAL: NCT03143231
Title: Normal Saline Versus Hypertonic Saline in the Treatment of Bronchiolitis
Brief Title: Normal Saline vs Hypertonic Saline in the Treatment of Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mariam Rajab, Chairperson of pediatrics department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1682016
Record Dates: First submitted 2017-04-21; First posted 2017-05-08 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Length of Hospital Stay
MeSH Terms: interventions — Saline Solution; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline (Experimental): Sodium Chloride 0.9% will be provided
  Interventions: Other: Normal saline
- Hypertonic saline (Experimental): 500 ml Sodium Chloride 0.9% with 60 ml Sodium Chloride 20% will be provided
  Interventions: Other: Hypertonic saline

INTERVENTIONS:
Other: Normal saline — The normal saline will be divided in 3ml aliquots that will be preserved in the pharmacy refrigerator between 2 and 60[0]C. Once a patient had been randomized, 6 aliquots would be prepared daily until the end of the trial.
  Arms: Normal saline
Other: Hypertonic saline — The mixture (500 ml Sodium Chloride 0.9% with 60 ml Sodium chloride 20%) will be divided in 3ml aliquots that will be preserved in the pharmacy refrigerator between 2 and 60[0]C. Once a patient had been randomized, 6 aliquots would be prepared daily until the end of the trial.
  Arms: Hypertonic saline

SUMMARY:
Background: Bronchiolitis is one of the most common and costly respiratory diseases in infants and young children. Despite the high prevalence and morbidity of bronchiolitis, therapy remains controversial. Supportive care ensuring adequate hydration and oxygenation remains the cornerstone of therapy for these infants.

Over the past 2 decades, research on bronchiolitis management has explored the use of nebulized hypertonic saline that rehydrate the airway surface liquid and improve mucociliary clearance, as well as reduce airway edema.

Aim:The aim of this study is to investigate whether the addition of frequently nebulized hypertonic saline to standard therapy affects the length of stay (LOS) of moderately ill infants hospitalized with bronchiolitis.

DETAILED DESCRIPTION:
The investigators will conduct this prospective double blind randomized clinical trial by comparing between 2 groups of patients with bronchiolitis, first group will receive 3% hypertonic saline and second group will receive 0.9% saline.

Data collection includes:

Name, Age, Mode of delivery, Birth weight, Current weight, Number of sibling, Immunization record, Duration of breast feeding, past medical history including number of wheezy chest, pneumonia, Parents level of education, Presence of Asthma / Allergic rhinitis in family, Pets /Smoke at home)

Using the validated Respiratory Distress Assessment Instrument (RDAI) investigators will assign patients a score before and at the end of treatment.

To prepare 3% sodium chloride, the investigators will dilute 60 ml 20% sodium chloride injection with 500 ml normal saline (NSS) 0.9%.

Length of stay will be measured in both groups, to establish the efficacy of hypertonic saline in reducing length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Infants up to 24 months of age with diagnosis of acute bronchiolitis
* In accordance with 2006 American Academy of Pediatrics (AAP) definition of bronchiolitis,we did not limit to the first episode of wheeze
* Patients with the diagnosis of bronchiolitis

Exclusion Criteria:

* Chronic lung or heart disease (hemodynamically significant cardiac disease, chronic lung disease / bronchopulmonary dysplasia requiring diuretics or oxygen)
* Cystic fibrosis, trisomy 21, immunodeficiency / transplant recipient, neuromuscular disease

Ages: 15 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | an average of 5 days
  from date of admission to discharge date

SECONDARY OUTCOMES:
transfer to pediatric intensive care unit (PICU) | an average of 3 days
  admission to PICU
use of mechanical ventilator | an average of 3 days
  clinical worsening of patients requiring mechanical ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Rajab, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No